CLINICAL TRIAL: NCT00262379
Title: Multicenter Study, Randomized and Pragmatic, Comparing Two Therapeutic Strategies : Use or Non-use of Epoetin Beta in Patients Infected by Chronic Hepatitis C and Treated by Combination Therapy Peginterferon Alfa-2a Plus Ribavirin
Brief Title: Use or Non-use of Epoetin Beta in Patients Infected by Chronic Hepatitis C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP 2005-01
Record Dates: First submitted 2005-12-05; First posted 2005-12-06 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic hepatitis C; peginterferon; ribavirin; epoetin beta
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — epoetin beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (No Intervention): HCV treatment with peginterferon plus ribavirin during 48 weeks
- Groupb (Active Comparator): HCV treatment with peginterferon plus ribavirin during 48 weeks plus epoetin beta under anemia conditions
  Interventions: Drug: epoetin beta (NeoRecormon®)

INTERVENTIONS:
Drug: epoetin beta (NeoRecormon®) — • Prescription of the epoetin beta : when blood concentration of hemoglobin is lower or equal to 12 g/dL in male or lower or equal to 11 g/dL in female
  Other Names: NeoRecormon®
  Arms: Groupb

SUMMARY:
The purpose is to demonstrate a correction of anemia in hepatitis C virus treatment with peginterferon plus ribavirin.

DETAILED DESCRIPTION:
Show that the correction of anemia by epoetin beta (NeoRecormon®) able to maintain a optimal dose of ribavirin (Copegus®). The study compares two therapeutic strategies : use or non-use of epoetin beta (NeoRecormon®) in patients infected by chronic hepatitis C and treated by combination therapy Peginterferon alfa-2a (Pegasys®) plus ribavirin (Copegus®). The main judgement criteria are :

* Sustained Viral Response (Week 72)
* Viral Response at the End of Treatment (Week 48)
* Quality of life
* Cumulative dose of ribavirin from D0-W24 and from W24-W48 periods
* Clinical and biological tolerance

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years old or above
* Patient with French social security or other equivalent health assurance
* Patient with informed consent
* Serologic evidence of chronic hepatitis C by detectable anti-HCV antibodies
* Patient infected by HCV genotype 1, 4, 5 or 6
* Compensated liver disease (Child-Pugh ≤ 6)
* Negative urine or blood pregnancy test (for women of childbearing potential) documented within the 24-hour period prior the enrollment in the study
* All fertile males and females receiving ribavirin must have effective contraception during treatment and during the 6 following months
* Patient naive of treatment with installation of treatment by investigator following criteria for use Peginterferon alfa-2a (Pegasys) and ribavirin (Copegus)

Exclusion Criteria:

* Women with ongoing pregnancy or breast feeding
* Male partner of pregnancy woman
* Minor
* Major protected by French law for biomedical study
* Co-infection by HBV or HIV
* History or other evidence of decompensated liver disease or Child-Pugh score > 6
* Clinical or radiological evidence (abdominal ultrasound, CT scan or MRI) of hepatocellular carcinoma
* IFN or ribavirin at any previous time
* Patient who received an erythropoetin within 2 months before inclusion
* History of epilepsy (during the last 6 months)
* Chronic cardiac insufficiency (stage III or IV in classification from the New York Heart Association [NYHA])
* Not controlled portal hypertension
* Antecedents or risk of venous thrombosis
* Surgery within 3 months before inclusion
* Serum creatinine level >15 mg/mL (130µmol/L)
* Deficiency in vitamin B9 and/or B12 (suspected with macrocytosis > 105 µm3)
* Thrombocytosis (platelets > 500 000/mm3)
* Chronic inflammatory syndrome (CRP > 10 mg/L)
* Deficiency not corrected in iron :
* Ferritin blood level < 10 µg/L Or - Transferrin saturation coefficient < 20 %
* History of neoplasia (except basocellular epithelioma and cervical cancer)
* Contraindications to use epoetin beta or an excipient from molecule to study (urea, polysorbate 20, glycine, leucine, isoleucine, threonine, glutamic acid, phenylalanine, benzoic acid, benzyl alcohol)
* Absence of written informed consent
* Exclusion time for another biomedical study
* Patient with blood concentration of hemoglobin lower or equal to 12 g/dL for male or lower or equal to 11 g/dL for female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2005-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Sustained Viral Response (Week 72) | Week 72
  Actual Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Values up to Week 24 in the Post-treatment Follow-up Period

SECONDARY OUTCOMES:
• Viral Response at the End of Treatment (Week 48) | Week 48
  Actual Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Values up to Week 48
• Quality of life | D0, W4, W12, W24, W48, W72
  * Questionnaire HQLQ
  * Fatigue Severity Scale HQLQ questionnaire and Fatigue Severity Scale
• Cumulative dose of ribavirin from D0-W24 and from W24-W48 periods | D0, W4, W8, W12, W16, W20, W24, W28, W32, W36, W40, W44, W48
  • Cumulating dose of ribavirin during following periods D0-W24 and W24-W48
• Clinical and biological tolerance | D0, W4, W8, W12, W16, W20, W24, W28, W32, W36, W40, W44, W48, W52, W60, W72
  Up to 72 weeks, includes all serious and other adverse events that newly occurred or worsened after treatment with PegIFNα-2a, ribavirin or epoetin beta

CONTACTS AND LOCATIONS:
Overall Officials: Françoise Lunel-Fabiani, MD, PhD, Principal Investigator — UH Angers
Locations (37):
- France (37):
  - H Aix en Provence, Aix-en-Provence
  - UH Angers, Angers
  - H Avignon, Avignon
  - H Bourgoin-Jallieu, Bourgoin
  - UH Brest, Brest
  - UH Caen, Caen
  - H Châteauroux, Châteauroux
  - UH Clermont Ferrand, Clermont-Ferrand
  - H Corbeil-Essonnes, Corbeil-Essonnes
  - H Creil, Creil
  - H Créteil, Créteil
  - UH Dijon, Dijon
  - H Dreux, Dreux
  - H Freyming-Merlebach, Freyming-Merlebach
  - H Grasse, Grasse
  - UH Grenoble, Grenoble
  - H La Roche sur Yon, La Roche-sur-Yon
  - H Le Mans, Le Mans
  - UH Limoges, Limoges
  - UH Lyon, Lyon
  - H Saint-Joseph, Marseille
  - H Montauban, Montauban
  - H montélimar, Montélimar
  - UH Montpellier, Montpellier
  - UH Nantes, Nantes
  - H Orléans, Orléans
  - H Tenon, Paris
  - H saint-Antoine, Paris
  - H Pau, Pau
  - UH Poitiers, Poitiers
  - UH Rennes, Rennes
  - UH Rouen, Rouen
  - H Saint-Dizier, Saint-Dizier
  - Arnault Tzanck Institute, Saint-Laurent-du-Var
  - UH Toulouse, Toulouse
  - H Tourcoing, Tourcoing
  - UH Tours, Tours